CLINICAL TRIAL: NCT04241302
Title: Development of a Mobile-app Based Free Field Click Test Against Conventional Free Field Voice Test
Brief Title: Development of a Mobile App FFVT vs FFCT : A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Goh Liang Chye, Principal Investigator, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 52296
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Deafness
Keywords: Mobile App; Clinical trial; Audiology; Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Intervention Model Description: Free Field Voice test vs Free Field Click Test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Field Voice test (Active Comparator): The examiner will inform the patient to repeat a sequence of Spondee words or a combination of numbers and letters whispered by the examiner initially. The examiner will be standing at the same distances as in the FFCT examination (starting with 2 feet). If the patient fails to hear the whispered voice at 2 feet, the examiner increases the loudness of voice to conversational tone at the same distance. The test is repeated thrice each time with a different set of Spondee words to avoid the patients recognizing the same sequence. If the patient is unable to respond, the examiner moves closer to 6 inches and whispers to the patient, and if no further response, then, conversational voice is used. The patient's free-field threshold is the voice and distance level at which more than 50% correct is obtained.
  Interventions: Diagnostic Test: Pure Tone Audiogram
- Free Field Click Test (Experimental): The app is designed by our team by a broadband (500-3000 Hz) click sound of 30-40 dB for soft sound/whisper and 60-70dB for loud sound/conversation voice. This app is designed by the Flutter-Dart programming tool and the speaker is produced via hand-held devices of Apple and Android brands. The tone is produced 3 times, with 2 out of 3 answers are considered as the patient's hearing threshold. The examiner stands at the distance of 2 feet away behind the seated patient and a soft sound from the FFCT is tested. The patient is then asked to respond yes or to nod if able to hear the sound. When the patient is unable to answer or no response is received upon thrice testing, the examiner then moves closer to 6 inches to the patient and again the soft sound is tested thrice. Loud sound is then tested if the patient is unable to respond, starting from 2 feet distance for three times. And then, the loud sound is tested at 6 inches of distance if no further response is obtained.
  Interventions: Diagnostic Test: Pure Tone Audiogram

INTERVENTIONS:
Diagnostic Test: Pure Tone Audiogram — A Pure Tone Audiogram is done in a sound proof room in both cases of Free Field Voice Test and Free Field Click Tests to identify the Pure Tone Average (Hearing Threshold Average of 500Hz,1000Hz and 2000Hz).

SUMMARY:
This is an open-labelled randomised controlled trial involving 2 groups which are Free Field voice test vs Free Field Click tests using digital hand-held devices. This study will be done at a sound-proof room in ORL clinic in Hospital Sultanah Aminah, Johor, Malaysia from January till July 2020.

DETAILED DESCRIPTION:
This is an open-labelled randomized controlled trial involving 2 groups which are Free Field voice test vs Free Field Click test (digital hand-held device). There will be no follow up for these participants as it is a one off assessment in most cases. Participants from the Otolaryngology clinic of Hospital Sultanah Aminah Johor Bahru will initially be screened during office hours for suitability based on our inclusion and exclusion criteria. Participants whom are interested will then be counselled and a consent form will be provided to the participants and he/she will be given sufficient time to consider before providing a signature on the consent forms.

The app is designed by the investigators using a broadband (500-3000 Hz) click sound of 30-40 dB for soft sound/whisper and 60-70dB for loud sound/conversation voice. This app is designed by using the Flutter-Dart programming tool and the speaker is produced via hand-held devices of Apple and Android brands. The tone is produced 3 times, with 2 out of 3 answers are considered as the participant's hearing threshold. The investigators stands at the distance of 2 feet away behind the seated participant and a soft sound from the FFCT is tested. The participant is then asked to respond yes or to nod if able to hear the sound. When the participant is unable to answer or no response is received upon third testing, the examiner then moves closer to 6 inches to the participant and again the soft sound is tested thrice. Loud sound is then tested if the participant is unable to respond, starting from 2 feet distance for three times. And then, the loud sound is tested at 6 inches of distance if no further response is obtained.

The same is done for the group of participants randomised into the Free Field voice test group. The investigator will inform the participant to repeat a sequence of Spondees words or a combination of numbers and letters whispered by the examiner initially. The investigator will be standing at the same distances as in the Free Field Click test examination (starting with 2 feet). If the participant fails to hear the whispered voice at 2 feet, the investigator increases the loudness of voice to conversational tone at the same distance. The test is repeated thrice each time with a different set of Spondee words to avoid the participants from recognizing the same sequence. If the participant is unable to respond, the investigator moves closer to 6 inches and whispers to the participant, and if no further response, then, conversational voice is used. The participant's free-field threshold is the voice and distance level at which more than 50% correct is obtained.

Both the FFVT and FFCT tests are done in a sound-proof room or a reasonably quiet room. The investigator stands behind the participant throughout the examination to prevent any lip reading. Each ear is tested individually, starting with the better ear and the non-test ear is masked by the participant by either gently occluding the ear canal with a finger or by tragal rubbing. The other ear is assessed similarly. Expected duration for the completion of a FFVT or FFCT is estimated to be approximately 5-10 minutes depending on severity of hearing loss where-else the duration for a diagnostic PTA would take between 10-20 minutes depending on complexity of hearing loss. This is a standard procedure in PTA practice and no additional steps were undertaken specifically for the purpose of this study.

As this is a study to compare the sensitivity and specificity of FFVT and FFCT, the study end-point involves the subjective hearing threshold obtained from the participant upon hearing the tested sound. The subjective threshold is measured under 5 categories which is whispering sounds at 2 feet (from the participants), whispering sounds at 6 inches, Conversational sounds at 2 feet, Conversational sounds at 6 inches and finally not being able to hear at all. The measurements of the 2 groups will then be compared to the pure tone average obtained through pure tone audiogram.

ELIGIBILITY:
Inclusion Criteria:

i) Age 18-80 years old ii) Chief complaint of reduced hearing -unilaterally or bilaterally iii) Able to communicate with the examiners iv) Post-traumatic patients with uni/bilateral hearing loss

Exclusion Criteria:

i) Age < 18 or > 80 years old ii) Uncooperative patient iii) Not consented iv) Intellectually-challenged v) Pregnant ladies vi) Previous ear surgery/ear tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Subjective hearing threshold | 15 minutes
  To compare the sensitivity and specificity of FFVT and FFCT, the study end-point involves the subjective hearing threshold obtained from the patient upon hearing the tested sound and comparing results to Pure Tone Audiogram and obtaining the Pure Tone Average

SECONDARY OUTCOMES:
Gender comparison | 15 minutes
  Comparison of sensitivity of hearing threshold detection of both Free field Voice test and Free Field click test between genders
Age Comparison | 15 minutes
  Comparison of sensitivity of hearing threshold detection of both Free field Voice test and Free Field click test on different age groups
Tympanogram comparison | 15 minutes
  Comparison of sensitivity of hearing threshold detection of both Free field Voice test and Free Field click test when tested with a tympanogram device
Laterality comparison | 15 minutes
  Comparison of sensitivity of hearing threshold detection of both Free field Voice test and Free Field click test between unilateral and bilateral hearing loss

CONTACTS AND LOCATIONS:
Overall Officials: Goh Liang Chye, MS (ORL-HNS), Study Director — Otorhinolaryngologist; Thilaga Rajendren, MBBS, Principal Investigator — Medical officer
Locations (1):
- Hospital Sultanah Aminah Johor Bahru, Johor Bahru, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Pirozzo S, Papinczak T, Glasziou P. Whispered voice test for screening for hearing impairment in adults and children: systematic review. BMJ. 2003 Oct 25;327(7421):967. doi: 10.1136/bmj.327.7421.967. PMID 14576249
- [Result] Dempster JH, Mackenzie K. Clinical role of free-field voice tests in children. Clin Otolaryngol Allied Sci. 1992 Feb;17(1):54-6. doi: 10.1111/j.1365-2273.1992.tb00988.x. PMID 1555319
- [Result] McShefferty D, Whitmer WM, Swan IR, Akeroyd MA. The effect of experience on the sensitivity and specificity of the whispered voice test: a diagnostic accuracy study. BMJ Open. 2013 Apr 18;3(4):e002394. doi: 10.1136/bmjopen-2012-002394. Print 2013. PMID 23604349